CLINICAL TRIAL: NCT00407108
Title: Perfluorocarbon Perfused Vitrectomy and 3D Vitrectomy System in Advanced Diabetic Retinopathy
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APEC-005
Record Dates: First submitted 2006-06-30; First posted 2006-12-04 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Retinopathy
Keywords: vitreoretinal surgery
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Vitrectomy

INTERVENTIONS:
Procedure: Vitrectomy

SUMMARY:
To investigate the feasibility and advantages of using perfluorocarbon liquid (PCL) perfusion to remove vitreous during suction-cutting vitrectomy using a dual, dynamic drive (3D)technology. In complicated surgeries in advanced diabetic retinopathy and retinal detachment

ELIGIBILITY:
Inclusion Criteria:

* Advanced diabetic retinopathy with retinal detachment

Exclusion Criteria:

* Retinal detachments of more than 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2006-03 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Surgical time
Facility of surgical maneuvers

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Quiroz-Mercado, MD, Principal Investigator — Asociación para Evitar la Ceguera en México
Locations (1):
- Asociación para Evitar la Ceguera en Mexico, Hospital "Luis Sanchez Bulnes", Mexico City, Mexico DF, Mexico